CLINICAL TRIAL: NCT01059227
Title: Effects of a CRF1 Receptor Antagonist on Human Startle in Normal Female Volunteers
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100049; 10-M-0049
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2015-08-14

CONDITIONS: Anxiety Disorders
Keywords: Treatment; Anxiety; Fear; Fear Potentiated Startle; Healthy Volunteer; HV
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
Background:

- Research has shown that the hormone corticotropin-releasing hormone (CRH) is involved in stress and anxiety, and that drugs that block the effect of CRH in the body can reduce anxiety. GSK561679 is an experimental drug that attempts to reduce anxiety by blocking the effect of CRH. Researchers are interested in comparing GSK561679 with other treatments for anxiety.

Objectives:

- To determine the effectiveness of GSK561679 compared with placebo and alprazolam (Xanax), as a possible treatment for fear and anxiety.

Eligibility:

- Healthy female volunteers between 21 and 50 years of age.

Design:

* This study will involve one screening visit, four testing visits, and one follow-up visit over a period of 8-9 weeks. The testing sessions will be between 6-11 days apart.
* Participants must follow these dietary restrictions to participate in the study.
* No nicotine, alcohol, or caffeine (including chocolate and soft drinks) for 24 hours before the start of the study.
* No nicotine in the past 6 months, and no nicotine until the final blood sample is collected at the follow-up visit.
* No alcohol or caffeine for 24 hours before a testing visit or for 72 hours after each visit.
* No grapefruit or grapefruit products from 14 days before the first dose of study medication until collection of the final blood sample.
* Participants will receive a dose of GSK561679, alprazolam, or placebo 3 hours before the testing, and will take an additional pill 1 hour before the testing.
* During the tests, participants will receive brief electric shocks and hear sudden loud noises. The noises and shocks will be given over a period of approximately 40 minutes per session.
* Skin conduction, heart rate, and blinking will be monitored throughout the tests, and participants will be asked about anxiety levels and will be tested on mood, memory, and concentration. Blood and saliva samples will also be taken during these sessions.
* Participants will stay in the clinical center for 1 to 2 hours after the study testing to ensure that the sedation has worn off. Participants will not be allowed to drive home or take public transportation alone after study visits, so alternative transportation must be arranged.

DETAILED DESCRIPTION:
Objective: This proposal is a part of an integrated project to test the efficacy of a candidate anxiolytic, a CRF1 receptor antagonist, provided by GlaxoSmithKline (GSK) as part of The Emory-MSSM-GSK-NIMH Collaborative Mood Disorders Initiative, using fear-potentiated startle. The anti-fear and anxiolytic activity of a single dose of the highly specific CRF1 antagonist GSK561679 will be evaluated in healthy female subjects using models of phasic (fear) and sustained (anxiety) aversive states derived from humans and from pre-clinical studies in rodents.

Study population: The study population will consist of 30 healthy female volunteers, 21-50 years of age, and of diverse racial and ethnic backgrounds.

Design: The study will use a double-blind cross-over design in which each subject will receive placebo, Alprazolam (1 mg), and a low (50 mg) and high (400 mg) dose of GSK561679. We will examine the effect of these drugs on the potentiation of startle during anticipation of no-shock, predictable shock signaled by a discrete threat cue, and unpredictable shock.

Outcome measures: The main outcome measures are the magnitude of the startle reflex and retrospective anxiety during each condition. Secondary measures will include the skin conductance response and changes in heart rate, as well as measures of HPA activity.

ELIGIBILITY:
* INCLUSION CRITERIA:

HEALTHY FEMALE VOLUNTEERS as determined by a responsible physician, based on a medical evaluation including own and familial medical history, physical examination, psychiatric history, psychiatric evaluation, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.

Females between the ages of 21 and 50 who are free of current psychopathology and free of past psychopathology of mood and anxiety disorder, psychotic disorder, and substance drug addiction

Organic central nervous system disorders

Able to give consent

A negative urine toxicology

For females of child-bearing potential, negative pregnancy urine test

For females child-bearing potential, use of two effective birth control methods* for the duration of the study or abstinence.

Abstinence from ingesting nicotine for at least 6 months before the start of the study.

*See specific criterion for effective birth control methods listed below.

EXCLUSION CRITERIA:

Subjects with an unstable medical disorder or a disorder (including surgical interventions) that would likely interfere with the action, absorption, distribution, metabolism or excretion of GSK561679, may pose a safety concern, or interfere with accurate assessment of safety.

1. Lifetime or current diagnosis of schizophrenia or other psychotic disorder, mood or anxiety disorder, substance abuse in the last 12 months or lifetime dependence, alcohol abuse in the last 12 months or lifetime dependence. Current Axis I disorder. Clear evidence of a first-degree relative with history of psychosis, bipolar disorder or major depression as determined by the family history interview method; specifically, participant will know diagnosis or treatment in order to confirm presence of disorder.
2. Subject is currently participating in another clinical trial in which she is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month
3. Current evidence or history of significant unstable medical illness or organic brain impairment, including stroke, epilepsy, CNS tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, renal or hepatic impairment that would likely interfere with the action, absorption, distribution, metabolism, or excretion of GSK561679. Abnormal EKG.
4. DSM-IV substance abuse within the past year. Subject has a positive urine test for illegal drug use.
5. Diagnosis of anorexia nervosa or bulimia
6. Subject has a documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis (hepatitis B surface antigen and/or hepatitis C antibody), and/or clinically significant hepatic enzyme elevation including any one of the following enzymes greater than 1.5 times the upper limit of normal (ULN) value (ALT, AST, ALP, total or direct bil > 1.5 times the ULN, unless consistent with presumed or diagnosed Gilbert s disease
7. Subject has taken systemic corticosteroids within 2 weeks of the Randomization Visit
8. All prescription or non-prescription medications and herbal remedies are prohibited within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication and until completion of follow-up procedures, unless in the opinion of the investigator the medication will not interfere with the study procedures or compromise study safety, e.g. rescue medication. As an exception, acetaminophen, no more than 2g/day, and birth control pills are permitted during the study.
9. Subject who is likely to require the use of the following medications:

   * Chronic (for more than 2 weeks), regular NSAID use unless administered concomitantly with an anti-secretory agent (i.e. proton-pump inhibitor or histamine-2 receptor antagonist)
   * Any use of aspirin (including low dose)
10. Subject has taken non-psychoactive (prescription or non-prescription), dietary, or herbal products, with a narrow therapeutic index, that are metabolized via the cytochrome P450 3A4 or 2C9 pathway (warfarin), or transported via OATP1B1 or P-gp, within 2 weeks (or 5 half-lives, whichever is longer) prior to the Randomization Visit.
11. Subject has taken other (nonpsychoactive) prescription, nonprescription, dietary, or herbal products that are potent inducers or inhibitors of the cytochrome P450 3A4 pathway for 2 weeks (or 5 half lives, whichever is longer) prior to the Randomization Visit.
12. Subject has participated in a study with an investigational drug within the period of 30 days prior to screening for this study
13. Pregnancy or lactation*
14. Subjects who, in the opinion of the investigator, would be noncompliant with the visit schedule or study procedures (e.g. illiteracy, planned vacations, or planned hospitalizations during the study).
15. Any laboratory abnormality that in the investigator s judgment is considered to be clinically significant (blood pressure, ECG, TSH, LFT, etc.)
16. Previous treatment with CRF1 receptor antagonist
17. Allergy to benzodiazepines
18. Medical conditions that would influence psychophysiological responses (e.g., cardiovascular disease, previous myocardial infarction, angina, uncontrolled hypertension).
19. A history of peptic ulcer disease (PUD)

    * A serum pregnancy test is performed during the screening. Since this test might not detect the very early stage of pregnancy (i.e. maximum of 10 day period between fertilization and implantation), women of child-bearing age are excluded from the study if they do not use at least two effective birth control methods for 15 days prior to receiving the study drug. Acceptable methods of birth control include: a double-barrier method (condoms or diaphragm) combined with spermicide; hormonal contraceptives plus single barrier (birth control pills, implants [Norplant] or injections [Depo-Provera]), Intrauterine Device (IUD), or abstinence (no sexual activity).

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-01-22; Study Completion 2015-08-14

PRIMARY OUTCOMES:
Magnitude of the startle reflex | One year

SECONDARY OUTCOMES:
Skin conductance response and heart rate | One year

CONTACTS AND LOCATIONS:
Overall Officials: Christian Grillon, Ph.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baas JM, Grillon C, Bocker KB, Brack AA, Morgan CA 3rd, Kenemans JL, Verbaten MN. Benzodiazepines have no effect on fear-potentiated startle in humans. Psychopharmacology (Berl). 2002 May;161(3):233-47. doi: 10.1007/s00213-002-1011-8. Epub 2002 Mar 20. PMID 12021826
- [Background] Barlow DH. Unraveling the mysteries of anxiety and its disorders from the perspective of emotion theory. Am Psychol. 2000 Nov;55(11):1247-63. doi: 10.1037//0003-066x.55.11.1247. PMID 11280938
- [Background] Blanchard RJ, Yudko EB, Rodgers RJ, Blanchard DC. Defense system psychopharmacology: an ethological approach to the pharmacology of fear and anxiety. Behav Brain Res. 1993 Dec 20;58(1-2):155-65. doi: 10.1016/0166-4328(93)90100-5. PMID 7907880